CLINICAL TRIAL: NCT04447430
Title: Bright Light Therapy in Pregnant Women With Major Depressive Disorder: a Randomized, Double-blind, Placebo-Controlled Study
Brief Title: Light Therapy to Improve Symptoms in Pregnant Women With Major Depressive Disorder
Acronym: GZPHBLT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Psychiatric Hospital (Other Government)
Collaborators: The Third Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Kangguang Lin, Department of Affective Disorder, Guangzhou Psychiatric Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GuangzhouPHBLT
Record Dates: First submitted 2020-06-23; First posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Major Depressive Disorder
Keywords: Light therapy; Major Depressive Disorder; Pregnancy
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bright light group (Experimental): treat patients with bright light (10000 lux)
  Interventions: Device: bright light
- dim red light group (Placebo Comparator): treat patients with dim red light (100 lux)
  Interventions: Device: dim red light

INTERVENTIONS:
Device: bright light — treat patients with bright light, 30 min per day, 7 times per week, over 6 weeks
  Arms: bright light group
Device: dim red light — treat patients with dim red light, 30 min per day, 7 times per week, over 6 weeks
  Arms: dim red light group

SUMMARY:
This study will investigate the effectivenss of bright light therapy(10000 lux white)on pregnant women with major depression disorder.

DETAILED DESCRIPTION:
Depression during pregnancy is a common and high impact disease.Children who are exposed to maternal depression during pregnancy have a higher risk of adverse birth outcomes, such as low birth weight, and more often show cognitive, emotional and behavioral problems.Therefore, early detection and prompt treatment of depression during pregnancy can benefit both mother and child.However, the window of opportunity in pregnancy is small and from the perspective of the child postponement is in fact non-treatment. Psychotherapy might take a long time to be effective and do not work for all people. Further, the safety of pharmacological treatment for pregnant women with depression is still a big concern .Psychiatric medication use for depression in pregnancy may also pose a risk of fetal growth retardation and preterm delivery, as well as withdrawal symptoms in the new born. Therefore, investigating non-pharmacological approaches to treating depression during pregnancy is urgent and relevant, for both mother and child. Preliminary evidence shows that bright light therapy (BLT) is an effective treatment for pregnant women with depression based on several theoretical and clinical considerations, with effect size around 0.45 and without adverse effects to the new born. In this study we aim to investigate the effectiveness of BLT on pregnant women with major depression.

ELIGIBILITY:
Inclusion Criteria:

Women; 18~45 years of age; medically healthy, with normal ocular function; 13~28 weeks pregnancy; DSM-V diagnosis of major depressive disorder HAMD score ≥18

Exclusion Criteria:

DSM-V defined bipolar disorder、schizophrenia、schizoaffective disorder,anxiety disorders; substance Use Disorders; substance use within the last 6 months; suicidal ideation, suicidal attempt, suicide behavior, and attempted suicide; being treated by the light therapy; with antidepressant in recent 2 months; Multiple pregnancy; Any obstetrical care or medications for physical disorders that might confound treatment results; current use of β-adrenergic blockers, melatonin, or St. John's wort; thyroid function test results inconsistent with normal pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-06-12 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in depressive symptoms from baseline | Week2;Week6
  Depressive symptoms will be measured by Hamilton Depression Rating Scale (HAMD)

SECONDARY OUTCOMES:
Changes in anxious symptoms from baseline | week 2; week 6
  anxious symptoms will be measured by the Hamilton Anxiety Scale(HAMA)

CONTACTS AND LOCATIONS:
Overall Officials: Kangguang Lin, MD,PhD, Principal Investigator — Guangzhou Brain Hospital(Guangzhou Psychiatric Hospital)
Locations (1):
- Guangzhou Brain Hospital (Guangzhou Huiai Hospital), Guanzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No